CLINICAL TRIAL: NCT00895843
Title: Protective Analgesia Using Bupivacaine and Conventional Release Ibuprofen Versus Bupivacaine and Sustained Release Ibuprofen for Postoperative Pain Relief in Patients Undergoing Third Molar Surgery: a Randomised Controlled Trial
Brief Title: Protective Analgesia for Postoperative Pain Relief Following Day Case Oral Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Manchester University NHS Foundation Trust (Other Government)
Responsible Party: Professor Paul Coulthard, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 9938
Record Dates: First submitted 2009-03-24; First posted 2009-05-08 (Estimated); Results first posted 2009-05-08 (Estimated); Last update posted 2009-06-01 (Estimated); Status verified 2009-05

CONDITIONS: Postoperative Pain; Wisdom Tooth
Keywords: Third molar
MeSH Terms: conditions — Pain, Postoperative | interventions — Ibuprofen; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional ibuprofen (Active Comparator)
  Interventions: Drug: ibuprofen; Drug: Bupivacaine
- Brufen retard (Experimental)
  Interventions: Drug: Brufen retard; Drug: Bupivacaine

INTERVENTIONS:
Drug: Brufen retard — Single dose 2 x 800mg tablets 2 hours prior to surgery
  Other Names: sustained release ibuprofen; modified release ibuprofen
  Arms: Brufen retard
Drug: ibuprofen — Single dose ibuprofen 2 x 200mg tablets 2 hours prior to surgery
  Other Names: Brufen; neurofen; conventional release ibuprofen
  Arms: Conventional ibuprofen
Drug: Bupivacaine — Up to 10ml of Bupivacaine 0.5% with 1:200,000 Adrenaline given prior to surgical incision as inferior alveolar nerve block and long buccal nerve infiltration.
  Other Names: Marcain 0.5% with 1 in 200,000 epinephrine

SUMMARY:
The purpose of this study is to investigate whether robust analgesic regime (protective analgesia) can improve postoperative pain experience for patients undergoing lower wisdom teeth extraction under day case general anaesthetic.

DETAILED DESCRIPTION:
The aim of the study was to demonstrate and improve postoperative pain experience using protective analgesia for patients undergoing oral surgery under day case general anaesthesia.

The primary objective was to investigate the efficiency of protective analgesia using combined effects of sustained release ibuprofen and bupivacaine nerve block in attenuation of postoperative pain following impacted third molar surgery under day case general anaesthesia.

The secondary objective was to document the safety and tolerability profile of conventional release versus sustained released ibuprofen with bupivacaine block in subjects undergoing impacted third molar surgery under day case general anaesthesia.

ELIGIBILITY:
Inclusion Criteria:

* healthy male and female patients aged 18 years and over
* patients requiring removal of one or more third molars, with at lease one completely or partially impacted in the mandible needing bone removal

Exclusion Criteria:

* history of allergy to NSAIDs
* pregnant
* history of GI disease
* history of bleeding disorders
* alcohol dependancy
* drug abuse

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2006-11; Primary Completion 2007-12 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul Coulthard, BDS FDS PhD, Principal Investigator — University of Manchester
Locations (2):
- United Kingdom (2):
  - Central Manchester and Manchester Children's NHS University Hospitals, Manchester, Lancashire
  - Central Manchester NHS Foundation Trust, Manchester, Lancashire

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Conventional Ibuprofen | Brufen Retard
Started | 60 | 62
Completed | 48 | 50
Not Completed | 12 | 12
Not completed — Protocol Violation | 12 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Conventional Ibuprofen | Brufen Retard | Total
Number analyzed (Participants) | 60 | 62 | 122
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0.0
  Between 18 and 65 years | 60 | 62 | 122.0
  >=65 years | 0 | 0 | 0.0
Age Continuous [Mean (Standard Deviation); unit: years] | 28.71 (5.809) | 28.82 (6.262) | 28.77 (6.013)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 16 | 56.0
  Male | 20 | 46 | 66.0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 60 | 62 | 122.0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Needing Rescue Medication
Description: Number of patients who required rescue medication within 6 hours
Time Frame: At 6 hours
Measure: Number; unit: Participants
Arm/Group | Conventional Ibuprofen | Brufen Retard
Number analyzed (Participants) | 48 | 50
Participants | 32 | 29

2. Secondary Outcome: Mean Pain Intensity
Description: Mean VAS scores of pain intensity for each time points
Time Frame: 30 mins, 1 hour, 6 hours, 24 hours and 48 hours after surgery
Reporting Status: Not Posted
Measure: Mean (Full Range); unit: VAS pain score 0 to 100

3. Secondary Outcome: Time to Rescue
Description: Time taken for rescue medication requirement
Time Frame: Between 30mins and 48 hours
Reporting Status: Not Posted
Measure: Median (95% Confidence Interval); unit: Minutes

4. Secondary Outcome: Pain Control/Relief
Description: Patient satisfaction scores
Time Frame: 48 hours after surgery (end of study)
Reporting Status: Not Posted
Measure: Mean (Full Range); unit: Numerical satisfaction score 0 to 10

ADVERSE EVENTS:
Arm/Group | Conventional Ibuprofen | Brufen Retard

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes